CLINICAL TRIAL: NCT01703780
Title: The Prevalence and the Prognosis of Resistant Hypertension Ascertained With Systemic Investigation and Optimal Treatment With Antihypertensive Drugs
Brief Title: The Diagnosis and Treatment of Resistant Hypertension, the Prevalence and the Prognosis
Acronym: doublepres
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Huazhong University of Science and Technology (Other); Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, hui rutai, Director, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2011BAI11B04
Record Dates: First submitted 2012-10-07; First posted 2012-10-11 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, peripheral white blood cells, urine

GROUPS / COHORTS (3):
- resistant hypertension: blood pressure remaining above goal (< 140/90 mm Hg for the general population and < 130/80 mm Hg for patients with diabetes or renal disease) despite using optimal doses of 3 antihypertensive agents of different classes(including a diuretic) for half to one year.
- controllable hypertension: blood pressure can reach 130/80 mm Hg or less in half year by use of optimal dose of less than 3 antihypertensive agents of different classes
- healthy control: 1. Age>50 years old
  2. Blood pressure ≤ 120/80 mm Hg( 24-hour blood pressure monitor or home blood pressure measurement at 6-9 am and 5-8pm, twice)
  3. No cardiovascular diseases: coronary artery disease(coronary angiography or CTA), cerebrovascular diseases(history, MRI-Lacunar brain stem), Carotid ultrasound
  4. No peripheral angiopathy (ABI<0.9 or lower extremity vessels Doppler ultrasound)
  5. No major cardiovascular risk factors:
     1. Dyslipidemia
     2. Diabetes
     3. Smoke within one year

SUMMARY:
Hypertension is still one of the major preventable risk factor for cardiovascular as well as cerebrovascular diseases globally, including ischaemic heart disease, heart failure, and renal impairment. Despite knowledge on hypertension and the availability of effective antihypertensive medications have progressed dramatically in recent years, the rate of uncontrolled hypertension ( reached 90%) remains high in China[1]. Among those with uncontrolled hypertension，it has been reported that 8.9% in all individuals with hypertension, and 12.8% in the hypertensive drug-treated population[2] are attributed to resistant hypertension. Resistant hypertension has been defined by AHA as high blood pressure (BP) in spite of appropriate lifestyle interventions and treatment of three or more different types of antihypertensive drugs at optimal dose, including at least one diuretics[3,4] or achieving adequate BP control with optimal doses of 4 or more antihypertensive drugs.

At present, not many specifically designed prospective researches concerning resistant hypertension are available. The prevalence of resistant hypertension is not well established and most knowledge about resistant hypertension derives from cross-sectional analyses and clinical trials. The patients with resistant hypertension have been expected to have server target damage, and worse prognosis than those who are non-resistant, but not well established either in the literature[2].

The purpose of this study is to determine the prevalence of resistant hypertension ascertained with systemic investigation and optimal treatment with antihypertensive drugs in community populations and clinic as well as the prognosis among patients with resistant hypertension compared with those who are non-resistant.

DETAILED DESCRIPTION:
Hypertension is still one of the major preventable risk factor for cardiovascular as well as cerebrovascular diseases globally, including ischaemic heart disease, heart failure, and renal impairment. Despite knowledge on hypertension and the availability of effective antihypertensive medications have progressed dramatically in recent years, the rate of uncontrolled hypertension ( reached 90%) remains high in China[1]. Among those with uncontrolled hypertension，it has been reported that 8.9% in all individuals with hypertension, and 12.8% in the hypertensive drug-treated population[2] are attributed to resistant hypertension. Resistant hypertension has been defined by AHA as high blood pressure (BP) in spite of appropriate lifestyle interventions and treatment of three or more different types of antihypertensive drugs at optimal dose, including at least one diuretics[3,4] or achieving adequate BP control with optimal doses of 4 or more antihypertensive drugs.

At present, not many specifically designed prospective researches concerning resistant hypertension are available. The prevalence of resistant hypertension is not well established and most knowledge about resistant hypertension derives from cross-sectional analyses and clinical trials. The patients with resistant hypertension have been expected to have server target damage, and worse prognosis than those who are non-resistant, but not well established either in the literature[2].

The purpose of this study is to determine the prevalence of resistant hypertension ascertained with systemic investigation and optimal treatment with antihypertensive drugs in community populations and clinic as well as the prognosis among patients with resistant hypertension compared with those who are non-resistant.

Subjects：Total 9638 patients with hypertension were recruited on December 31 2015，50% from 5 communities screening, 50% from consecutive clinic hypertensive patients. The expected rate of resistant hypertension is 6% in hypertensive population.

Objectives:

1. True prevalence of resistant hypertension In order to obtain the true burden of resistant hypertension, a uniform definition of resistant hypertension were applied, AHA definition[4], "high blood pressure (BP) remained in spite of appropriate lifestyle interventions and treatment of three or more different types of antihypertensive drugs at optimal dose, including at least one diuretics or achieving adequate BP control with optimal doses of 4 or more antihypertensive drugs.

   1. To exclude pseudoresistant hypertension
   2. To avoid inaccurate measurement of blood pressure
   3. To make sure that both the patients and the physicians are adherent to therapeutic plans and to lifestyle interventions.The physicians comply with guidelines and actively pursue adequate blood pressure for their patients. Ninety per cent of the patients take recommended optimal daily doses of their antihypertensive medications at follow-up for 6 months as well as more than 85% for 2 years(less than 50% at present) Incidence of resistant hypertension TREATMENT RECOMMENDATIONS This is a practical clinical trial,no specific antihypertensive drugs are going to be tested in the trial.The antihypertensive drugs are selected according to guidelines.

      Treatment duration: six months of intensive treatment(optimal dose and type of drugs),blood pressure does not reach goal.

      The treatment of secondary causes of hypertension are referred to pertinent specialists.

      Appropriate lifestyle interventions are always encouraged:

      Nonpharmacological therapy:

      Reversal of lifestyle factors contributing to treatment resistance,
      * DASH diet is encouraged to follow, lower salt diet (ideal goal< 100 mEq of sodium/24 h,evaluated with 24h urine collection), low fat and high fibre diet,
      * weight loss if obese or overweight,
      * moderation of alcohol intake to no more than two drinks per day for men and one drink for women or lighter-weight persons,
      * smoking cessation,
      * regular physical activity.

      Optimal pharmacological therapy

      Drug treatment of resistant hypertension:
      * Diuretics: Usually taking thiazide, among patients with an estimated glomerular filtration < 40 mL/min per m2(body surface area), thiazide diuretics become less effective and loop diuretics should be used instead, such as furosemide, which needs at least twice daily dosing due to its short half-life.
      * Aldosterone antagonists, add-on therapy to use in resistant hypertension: spironolactone 25 mg once a day.
      * In order to get better adherence to antihypertensive drug therapy, and better antihypertensive effects and less side effects, combination medicine is encouraged to use and the use of which class combinations follows guidelines and ASH recommendation(2011),but this is the choice of patients and physicians.
      * Renal denervation with catheter-based radiofrequency ablation is not performed in this trial.
   4. To rule out white-coat effect：It has been reported that 20%-30% of patients with apparent resistant hypertension referred for ambulatory BP monitoring in fact have normal BP readings[5].When patients have higher BP levels than 140 over 90 mmHg when measured by the physician than when assessed at home or with AMBP( ambulatory monitoring blood pressure) which is called white-coat hypertension. The patients with white-coat hypertension have less severe target organ damage and cardiovascular risk than those with persistent elevated blood pressure in ambulatory monitoring.
   5. Reversing of contributing lifestyle factors for high blood pressure.

      * Obesity
      * High dietary salt intake (controlled at 6 grams daily as possible as we can).
      * The recognition and avoid of other common contributing factors such as non-steroidal anti-inflammatory drug use, oral contraceptive hormones
      * The recognition and treatment of progressive renal impairment.
   6. To rule out carefully the potential reversible causes of hypertension by medical history, physical examination, biochemical evaluation, and/ or non-invasive imaging. If diagnosed， pertinent therapy is given to the secondary hypertension:

      * Sleep apnoea
      * Primary aldosteronism , reported prevalence of approximately 20% in resistant hypertension[6]
      * Renal parenchymal disease and renal artery stenosis
      * Aortic coarctation
      * Cushing syndrome
      * Pheochromocytoma
   7. Biochemical evaluation, including serum sodium, potassium, glucose, and creatinine (creatinine clearance); plasma aldosterone and renin activity.
   8. 24-h urine collection to estimate dietary sodium, potassium, and aldosterone excretion. Testing for urinary or plasma metanephrines/catecholamines is indicated only when pheochromocytoma is suspected
   9. Non-invasive imaging is mandatory when there is a suspicion of renal artery stenosis, adrenal adenoma/tumour, parenchymal renal disease or aortic coarctation
2. Target damage of resistant hypertension:

   1. left ventricular hypertrophy: ECG and echocardiography
   2. periphery artery disease: ABI,carotid
   3. kidney function: urinary microalbumin,cystatin C,creatinine eGFR
   4. coronary heart disease
   5. Stroke
3. Prognosis: hard endpoints: acute coronary syndrome (including unstable angina, fatal and non-fatal myocardial infarction), stroke,all cause death, cardiovascular death

Major modifications as follows:

1. Recruitment status: total 9638 patients with hypertension were recruited on July 31，2015. In order to observe the treatment resistance, more than 6 month-treatment period needed, so the recruiting was postponed to December 31, 2015, and treated-resistant hypertensives were diagnosed after full-dose antihypertensive treattment for 6 months or more(to December 31,2015).
2. Target Follow-Up Duration: according to the modified protocol by PI and scientific committee of the study, and approved by ethic committee, this study has been divided as two stages:

   Stage-1: study the prevalence of treated-resistant hypertension, to December 31 2015.

   Stage-2: follow up was extended for 3 years to investigate the association of genetic risk factors as well as pharmacoepigenomic changes in antihypertensive drug-related metabolism enzymes and drug receptors with clinical phenotypes, including primary clinical endpoints, total death, cardiovascular death, acute myocardial infarction, stroke; secondary clinical events: rate of resistant hypertension, target organ damage, left ventricular hypertrophy, chronic kidney disease.Financial funding was supported by Qingdao HuangHai pharmaceutical.co., LTD.
3. Intervention

Since this is practical clinical trial, patients were allowed to receive any following antihypertensive drugs and dosage adjustment was based on JNC-cited clinical trials and also the recommendation in JAMA[7].

* Angiotensin converting enzyme inhibitors: Captopril, Benazepril, Enalapril, Perindopril, Lisinopril
* Angiotensin II receptor antagonists: Candesartan Cilexetil, Valsartan, Telmisartan, Irbesartan, and Olmesartan
* β-blockers：Atenolol, Metoprolol，Bisolol
* Calcium channel blockers: Nifedipine, Amlodipine
* Diuretics: Hydrochlorothiazide, Indapamide

Treatment-Resistant Hypertension was defined as that blood pressure was still over 140/or over 90 mm Hg after taking 3 different classes of antihypertensive drugs for 6 months or more than 6 months, including one diuretics such as hydrochlorothiazide or indapamide or taking 4 or more than 4 different classes of antihypertensive drugs.

At stage-1 study, we investigated the prevalence of treated-resistant hypertension. But, the mechanism of treated-resistant hypertension has not been clarified. Previous study showed that a total of 248 drug metabolism pathways with known CYP involvement. Of 57 putatively functional human CYPs only about a dozen enzymes, belonging to the CYP1, 2, and 3 families, are responsible for the biotransformation of most foreign substances including 70%-80% of all drugs in clinical use[8]. We hypothesized that the resistance results from the either epigenomical modifications of the gene encoding the enzymes related to drug metabolism and the gene encoding drug receptors or genomic variants for cardiovascular disease (GWAS studies provided).

To test our hypothesis, we proposed the epigenomic-modified targets as DNA methylation of the gene encoding metabolism enzymes and receptors of antihypertensive drugs. Target-1 is CYP2D6, involved in quarter of total clinical used drug metabolism，40% of them are used to treat cardiovascular disease. Other important CYP 450 enzymes targets involved in cardiovascular drug metabolism are CYP3A family, CYP2C family[8].

For epigenomic study, patients were allowed to receive any one of the follow antihypertensive drugs and dosage adjustment was based on the JNC-7 cited clinical trials and the recommendation in JAMA[7]. The following antihypertensive therapy was used.

* Angiotensin converting enzyme inhibitors: Captopril, Benazepril, Enalapril, Perindopril, Lisinopril.
* Angiotensin II receptor antagonists: Candesartan Cilexetil, Valsartan, Telmisartan, Irbesartan, and Olmesartan.
* β-blockers：Atenolol, Metoprolol，Bisolol.
* Calcium channel blockers: Nifedipine, Amlodipine.
* Diuretics: Hydrochlorothiazide, Indapamide.

Sample：Peripheral white blood cells.

Sample collection：Before antihypertensive drugs, as well as year 1, 2, 3 on antihypertensive drug therapy (Time series with non-equivalent control group designs（multiple time series design).

ELIGIBILITY:
Inclusion Criteria:

Resistant hypertension,ascertained according to AHA criteria: blood pressure remaining above goal (< 140/90 mm Hg for the general population and < 130/80 mm Hg for patients with diabetes or renal disease) despite using optimal doses of 3 antihypertensive agents of different classes(including a diuretic) for half to one year.

controllable hypertension blood pressure can reach 130/80 mm Hg or less in half year by use of optimal dose of less than 3 antihypertensive agents of different classes

healthy control

* Age>50 years old
* Blood pressure ≤ 120/80 mm Hg( 24-hour blood pressure monitor or home blood pressure measurement at 6-9 am and 5-8pm, twice)
* No cardiovascular diseases: coronary artery disease(coronary angiography or CTA), cerebrovascular diseases(history, MRI-Lacunar brain stem), Carotid ultrasound
* No peripheral angiopathy (ABI<0.9 or lower extremity vessels Doppler ultrasound)
* No major cardiovascular risk factors: Dyslipidemia, Diabetes,Smoking within one year.

Exclusion Criteria:

* severe hepatic diseases
* mental diseases
* cancer
* systemic diseases

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50% hypertensive patients from community population, 50% hypertensive patients from clinic as consecutive patients
Sampling Method: Probability Sample
Enrollment: 9638 (Actual)
Dates: Start 2012-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Acute myocardial infarction | 3 years

SECONDARY OUTCOMES:
Stroke | 3 years
  ischemic stroke, hemorrhage stroke

OTHER OUTCOMES:
All cause death | 3 years
Cardiovascular death | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rutai Hui, MD & PhD, Principal Investigator — Cardiovascular Institute and Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical college
Locations (18):
- China (18):
  - FuWai Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The general hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital of southern medical university, Guangzhou, Guangdong
  - Hongxinglong Center Hospital, Shuangyashan, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - TongJi Hospital, TongJi Medical Colleage, HuaZhong University of Science and Technology, Wuhan, Hubei
  - The Third People's Hospital of Xuzhou, Xuzhou, Jiangsu
  - The First Bethun Hospital of Jilin University, Changchun, Jilin
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Rizhao Port Hospital, Rizhao, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The fourth military medical university, Xi’an, Shanxi
  - West China Hospital，Sichuan Univer, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Background] Gu D, Reynolds K, Wu X, Chen J, Duan X, Muntner P, Huang G, Reynolds RF, Su S, Whelton PK, He J; InterASIA Collaborative Group. The International Collaborative Study of Cardiovascular Disease in ASIA. Prevalence, awareness, treatment, and control of hypertension in china. Hypertension. 2002 Dec;40(6):920-7. doi: 10.1161/01.hyp.0000040263.94619.d5. PMID 12468580
- [Background] Persell SD. Prevalence of resistant hypertension in the United States, 2003-2008. Hypertension. 2011 Jun;57(6):1076-80. doi: 10.1161/HYPERTENSIONAHA.111.170308. Epub 2011 Apr 18. PMID 21502568
- [Background] Mansia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Struijker Boudier HA, Zanchetti A; European Society of Hypertension; European Society of Cardiology. 2007 ESH-ESC Guidelines for the management of arterial hypertension: the task force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). Blood Press. 2007;16(3):135-232. doi: 10.1080/08037050701461084. No abstract available. PMID 17846925
- [Background] Calhoun DA, Jones D, Textor S, Goff DC, Murphy TP, Toto RD, White A, Cushman WC, White W, Sica D, Ferdinand K, Giles TD, Falkner B, Carey RM; American Heart Association Professional Education Committee. Resistant hypertension: diagnosis, evaluation, and treatment: a scientific statement from the American Heart Association Professional Education Committee of the Council for High Blood Pressure Research. Circulation. 2008 Jun 24;117(25):e510-26. doi: 10.1161/CIRCULATIONAHA.108.189141. PMID 18574054
- [Background] Brown MA, Buddle ML, Martin A. Is resistant hypertension really resistant? Am J Hypertens. 2001 Dec;14(12):1263-9. doi: 10.1016/s0895-7061(01)02193-8. PMID 11775136
- [Background] Calhoun DA, Nishizaka MK, Zaman MA, Thakkar RB, Weissmann P. Hyperaldosteronism among black and white subjects with resistant hypertension. Hypertension. 2002 Dec;40(6):892-6. doi: 10.1161/01.hyp.0000040261.30455.b6. PMID 12468575
- [Background] Vongpatanasin W. Resistant hypertension: a review of diagnosis and management. JAMA. 2014 Jun 4;311(21):2216-24. doi: 10.1001/jama.2014.5180. PMID 24893089
- [Background] Zanger UM, Schwab M. Cytochrome P450 enzymes in drug metabolism: regulation of gene expression, enzyme activities, and impact of genetic variation. Pharmacol Ther. 2013 Apr;138(1):103-41. doi: 10.1016/j.pharmthera.2012.12.007. Epub 2013 Jan 16. PMID 23333322